CLINICAL TRIAL: NCT03850808
Title: The Incidence of Left Ventricular Dysfunction Following Pacemaker Placement: Differential Effects of Intrinsic AV Node Disease v. AV Node Ablation.
Brief Title: LV Dysfunction Following Pacemaker Placement
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Charles Henrikson, MD, Associate Professor of Medicine, Oregon Health and Science University
Other Study IDs: PPMLV-9879
Record Dates: First submitted 2013-09-25; First posted 2019-02-22 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: heart failure; permanent pacemaker; AV node dysfunction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- decline in left ventricular function: This group will be patients in whom a decline in left ventricular systolic function was found.
- preserved left ventricular function: This group will consist of patients in whom left ventricular systolic function is preserved.

SUMMARY:
Several studies have confirmed the link between chronic RV apical pacing and the development of heart failure and LV systolic dysfunction in some patients 1,2. However, questions continue to remain unanswered in regard to the adverse effects of RV pacing such as the exact amount of RV pacing that is detrimental to cardiac function and which subsets of patients are most at risk for developing cardiac dysfunction from chronic RV pacing. Rates of permanent pacemaker implantation have been increased over the last twenty years with expanding indications to include permanent pacing after AV node ablation for the treatment of drug refractory atrial fibrillation and other atrial tachy-arrhythmias. The current standard of practice is to minimize RV pacing however in patients that have had an AV node ablation right ventricular pacing cannot be avoided therefore it is important to identify if this particular group of patients is at an increased risk for developing worsening cardiac function. The purpose of this study is to compare cardiac function over time between patients that have undergone AV node ablation versus patients that have had pacemaker implantation for AV node dysfunction.

DETAILED DESCRIPTION:
Study Design This is a retrospective chart review of patients that have undergone permanent pacemaker implantation by the electrophysiology group at Oregon Health and Sciences University Hospital during the period between 01/2003 and 01/2013 for chronic RV pacing after AV node ablation or for AV node dysfunction.

Goal The goal of this study is to determine if patients requiring RV pacing after AV nodal ablation are at increased risk for developing worsening cardiac function secondary to chronic RV pacing compared to patients requiring RV pacing for AV node dysfunction.

Specific Objectives

* To determine the number of patients that have a permanent pacemaker implanted after AV node ablation and for AV node dysfunction within the last 10 years at OHSU Hospital.
* To determine the number of patients that have a biventricular pacemaker implanted with or without an implantable cardiac defibrillator within the last 10 years at OHSU Hospital (control group).
* Amongst those patients identified determine (1) left ventricular ejection fraction prior to permanent pacemaker or biventricular pacemaker implantation and over time (2) left ventricular volume and/or diameter prior to permanent pacemaker placement and over time (3) all cause mortality
* Amongst those patients identified determine incidence of new onset atrial fibrillation after permanent pacemaker or biventricular pacemaker implantation
* Amongst those patients identified determine incidence of inpatient admission of heart failure exacerbation defined as presenting symptoms of dyspnea, orthopnea, paroxysmal nocturnal dyspnea, increased lower extremity edema requiring IV diuretics

Methods

This is a retrospective chart review of patients that have undergone permanent pacemaker medical record system used at OHSU Hospital) with the help of an EPIC representative. If the patient was referred for permanent pacemaker or biventricular pacemaker implantation from a physician or medical group outside of OHSU records will be requested from that physician or medical group.

ELIGIBILITY:
Inclusion Criteria: Patients who have undergone permanent pacemaker placement for AV node dysfunction.

-

Exclusion Criteria: retrospective--n/a

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undergone permanent pacemaker placement for AV node dysfunction
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-09; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Systolic Function | 3 month and 1 year followup, if available (this is a chart review)
  This is a chart review to see if left ventricular systolic function changed after placement of a permanent pacemaker. Changed is defined as 10 percentage points of left ventricular ejection fraction.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Henrikson, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States